CLINICAL TRIAL: NCT05314023
Title: A Phase 3 Open-Label Immunogenicity and Safety Study of 2-Dose Regimens of V503, a 9-Valent Human Papillomavirus (HPV) Vaccine in Chinese Males 9 Through 14 Years Old and 3-Dose Regimen of V503 in Chinese Males 9 Through 19 Years Old
Brief Title: Immunogenicity and Safety of V503 in Chinese Males 9 Through 19 Years Old (V503-053)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-053; V503-053 (Other: Merck)
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Genital Warts
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 9 to 19 Years Old: Day 1, Months 2 and 6 (Experimental): Chinese males 9 to 19 years old will receive a 0.5 mL intramuscular (IM) injection of 9-valent HPV (9vHPV) vaccine on Day 1, Month 2 and Month 6
  Interventions: Biological: 9vHPV vaccine
- 9 to 14 Years Old: Day 1, and Month 6 (Experimental): Chinese males 9 to 14 years old will receive a 0.5 mL IM injection of 9vHPV vaccine on Day 1 and Month 6
  Interventions: Biological: 9vHPV vaccine
- 9 to 14 Years Old: Day 1 and Month 12 (Experimental): Chinese males 9 to 14 years old will receive a 0.5 mL IM injection of 9vHPV vaccine on Day 1 and Month 12
  Interventions: Biological: 9vHPV vaccine

INTERVENTIONS:
Biological: 9vHPV vaccine — A 9-valent HPV vaccine (Types 6, 11, 16, 18, 31, 33, 45, 52, and 58) will be administered as a 0.5 mL IM injection.
  Other Names: V503; GARDASIL™9

SUMMARY:
This study is designed to demonstrate non-inferior immunogenicity of 3 doses of the 9-Valent Human Papillomavirus (9vHPV) vaccine (GARDASIL™9, V503) in Chinese males 9 through 19 years of age, and 2 doses of the 9vHPV vaccine in Chinese males 9 through 14 years of age, compared to the 3 dose regimen in Chinese males 20 through 26 years of age (from Merck Protocol V503-052). The primary hypothesis is that each of the 3-dose regimen in Chinese males aged 9 through 19 years and 2-dose regimens in Chinese males aged 9 through 14 years induces non-inferior competitive Luminex immunoassay (cLIA) geometric mean titers (GMTs) at one month post last dose compared to the 3-dose regimen in Chinese adult males aged 20 through 26 years. A noninferiority margin of 0.67 in the GMT ratio (9 through 19 years of age or 9 through 14 years of age vs 20 through 26 years of age) is used for each HPV type.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy Chinese male.
* Has not had sexual debut at the time of enrollment, and does not plan on becoming sexually active during the vaccination period (Day 1 through one month post last dose).

Exclusion Criteria:

* Has a history of known prior vaccination with an HPV vaccine.
* Has a history of HPV-related external genital lesions, HPV-related intra-anal lesions, or HPV-related head and neck cancer.
* Has a history of severe allergic reaction that required medical intervention.
* Has received immune globulin or blood-derived products in the past 6 months or plans to receive any before one month post last dose.
* Has a history of splenectomy, is currently immunocompromised, or has been diagnosed with immunodeficiency, human immunodeficiency virus (HIV), lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition.
* Has received immunosuppressive therapy in the past year, excluding inhaled, nasal, or topical corticosteroids and certain regimens of systemic corticosteroids.
* Has a known thrombocytopenia or coagulation disorder that would contraindicate IM injections.

Ages: 9 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Chinese males only
Enrollment: 1590 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2029-02-19 (Estimated); Study Completion 2029-02-19 (Estimated)

PRIMARY OUTCOMES:
Competitive Luminex immunoassay (cLIA) GMTs to 9 vaccine types of 9vHPV vaccine at one month post last dose | Up to Month 13
  cLIA GMT to each of 9 vaccine types of 9vHPV vaccine at one month post last dose. The GMT for each HPV type will be reported in mMU/mL.
cLIA GMTs to 9 vaccine types of 9vHPV vaccine up to 60 months post last dose | Up to 72 months
  cLIA GMT to each of 9 vaccine types of 9vHPV vaccine at up to 60 months post last dose. The GMT for each HPV type will be reported in mMU/mL.
cLIA seropositivity percentages to 9 vaccine types of 9vHPV vaccine | Up to 72 months
  cLIA seropositivity to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.

SECONDARY OUTCOMES:
cLIA seroconversion percentages to 9 vaccine types of 9vHPV vaccine | Up to Month 13
  cLIA seroconversion to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.
Immunoglobulin G Luminex immunoassay (IgG LIA) GMTs to 9 vaccine types of 9vHPV vaccine at one month post last dose | Up to Month 13
  IgG LIA GMT to each of 9 vaccine types of 9vHPV vaccine at one month post last dose. The GMT for each HPV type will be reported in mMU/mL.
IgG LIA seroconversion percentages to 9 vaccine types of 9vHPV vaccine | Up to Month 13
  IgG LIA seroconversion to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.
Percentage of participants experiencing solicited injection-site adverse events (AEs), | Day 1 through Day 8 following any study vaccination
  An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Solicited injection-site AEs such as erythema, swelling, pain, and induration at the injection site will be recorded.
Percentage of participants experiencing solicited systemic AEs | Day 1 through Day 8 following any study vaccination
  An AE is any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Systemic AEs are those not categorized as injection-site AEs.
Percentage of participants experiencing serious AEs (SAEs) | Up to 72 months
  A SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
IgG LIA GMTs to 9 vaccine types of 9vHPV vaccine up to 60 months post last dose | Up to 72 months
  IgG LIA GMT to each of 9 vaccine types of 9vHPV vaccine up to 60 months post last dose. The GMT for each HPV type will be reported in mMU/mL.
IgG LIA seropositivity percentages to 9 vaccine types of 9vHPV vaccine | Up to 72 months
  IgG LIA seropositivity to each of 9 vaccine types of 9vHPV vaccine. The percentage of participants who are seropositive for each HPV type will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- China (5):
  - Liucheng County Centers for Disease Control and Prevention ( Site 0005), Liuchow, Guangxi
  - Center for Disease Control and Prevention of Rong An ( Site 0006), Liuchow, Guangxi
  - Loudi Public Health Hospital (Loudi Occupational Disease Prevention And Treatment Hospital) ( Site 0, Louxing District, Hunan
  - Yuechi Disease Prevention and Control Center ( Site 0002), Guang’an, Sichuan
  - Santai County Center for Disease Control and Prevention ( Site 0001), Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php